CLINICAL TRIAL: NCT03782896
Title: The Effects of Anesthetics on Persistent Pain Following Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC2018-09-029-003
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Chronic Post-Procedural Pain
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mastectomy group: All patients who received the mastectomy (breast conserving surgery and sentinel lymph node dissection)
  Interventions: Other: acute postoperative pain

INTERVENTIONS:
Other: acute postoperative pain — All patients assessed postoperative pain score in the recovery room and postoperative 2 month

SUMMARY:
Persistent postoperative pain occurs up to 25 to 60 % after mastectomy. This occurs at a higher frequency than the rate of invasive surgery.Therefore, many ways have been tried to study risk factors. A study was conducted to predict postoperative pain for items (preoperative pain, sensitivity, pain prediction). As a result, it was reported that the scope of surgery, pre-operative pain, young age, and depression were associated with persistent pain.

This study try to find out whether persistent pain after mastectomy is affected anesthetic factors appropriate anesthesia depth and opioid using standardized monitoring devices limited to similar surgical ranges.

DETAILED DESCRIPTION:
Persistent postoperative pain occurs up to 25 to 60 % after mastectomy. This occurs at a higher frequency than the rate of invasive surgery.Therefore, many ways have been tried to study risk factors. A study was conducted to predict postoperative pain for items (preoperative pain, sensitivity, pain prediction). As a result, it was reported that the scope of surgery, pre-operative pain, young age, and depression were associated with persistent pain.

There were reports of no association with anesthesia in the area of anesthesia to the high pain control requirement in the postoperative recovery room, 24 hours of high pain medication, use of inhalation agent, and a high dosage of remifentanil. However, an anesthesia-related study was either a retrospective study or anesthetic was injected with more than a clinical dose in order to make the difference following methods.

In this study, bispectral index is used to maintain anesthesia depth. In addition, the commercially available noninvasive pain depth equipment (Surgical Pleth Index) is used to assess the nociception-antinociception balance. Displays the automatically calculated values of SPI=100-(0.3*heartbeat interval + 0.7*photoplethysmographic pulse wave ampule) using a waveform with peripheral oxygen saturation. Through this process, patients want to objectify the amount of anesthetic agent used during surgery. And all patients are inserted the laryngeal mask airway.

This study would try find out whether persistent pain after mastectomy is affected anesthetic factors appropriate anesthesia depth and opioid using standardized monitoring devices limited to similar surgical ranges.

The investigators hypothesize that patients who suffered severe acute postoperative pain, regardless of their anesthesia method, have a higher incidence of persistent post-mastectomy pain.

ELIGIBILITY:
Inclusion Criteria:

-undergoing breast conserving surgery + sentinel lymph node dissection

Exclusion Criteria:

* cardiac arrythmia
* allergic history for drugs
* renal failure (Cr> 1.5 mg/dl)
* performing axillary lymph node dissection or Total mastectomy
* difficult airway and failed to place laryngeal mask airway properly

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the 20-70 year old patients who undergoing breast conserving surgery + sentinel lymph node dissection at samsung medical center
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
persistent pain | postoperative 2 months
  persistent postoperative pain after mastectomy (Numeric rating pain score (NSR: no pain=1, worst pain=10)
acute postoperative pain | postoperative 1 hour
  acute postoperative pain in the recovery room measured by Numeric rating pain score (NSR: no pain=1, worst pain=10)

SECONDARY OUTCOMES:
inhalation agent | intraoperative
  inhalation anesthetics use or total intravenous anesthesia
opioid consumption | intraoperative
  the amount of opioid
surgical anxiety level | 1 day before surgery
  (0: not anxiety-100: extremely anxious)
anticipate pain | 1 day before surgery
  (0: no pain-100: a bad as you can imagine)
anticipated pain medication need | 1 day before surgery
  (0: none at all, 1: much less than average, 2: less than average, 3: average, 4: more than average, 5: much more than average)
surgery factor | intraoperative
  the incision size and the number of excision of lymph node
The surgical pleth index | intraoperative
  the highest surgical pleth index score in time of start anesthesia and ene of anesthesia
The pain score of discharge | on the 1 day of discharge
  Numeric rating pain score (NSR: no pain=1, worst pain=10)
the consumption of postoperative analgesia | postoperative 72 hours
  the consumption of postoperative analgesia during in-hospital day

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schreiber KL, Martel MO, Shnol H, Shaffer JR, Greco C, Viray N, Taylor LN, McLaughlin M, Brufsky A, Ahrendt G, Bovbjerg D, Edwards RR, Belfer I. Persistent pain in postmastectomy patients: comparison of psychophysical, medical, surgical, and psychosocial characteristics between patients with and without pain. Pain. 2013 May;154(5):660-668. doi: 10.1016/j.pain.2012.11.015. Epub 2012 Dec 5. PMID 23290256
- [Background] Cui L, Fan P, Qiu C, Hong Y. Single institution analysis of incidence and risk factors for post-mastectomy pain syndrome. Sci Rep. 2018 Jul 31;8(1):11494. doi: 10.1038/s41598-018-29946-x. PMID 30065342
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Pan PH, Tonidandel AM, Aschenbrenner CA, Houle TT, Harris LC, Eisenach JC. Predicting acute pain after cesarean delivery using three simple questions. Anesthesiology. 2013 May;118(5):1170-9. doi: 10.1097/ALN.0b013e31828e156f. PMID 23485992
- [Background] Lefebvre-Kuntz D, Duale C, Albi-Feldzer A, Nougarede B, Falewee MN, Ouchchane L, Soule-Sonneville S, Bonneau J, Dubray C, Schoeffler P. General anaesthetic agents do not influence persistent pain after breast cancer surgery: A prospective nationwide cohort study. Eur J Anaesthesiol. 2015 Oct;32(10):697-704. doi: 10.1097/EJA.0000000000000215. PMID 26053994